CLINICAL TRIAL: NCT03554330
Title: The Combined Use of Radiofrequency-catheter-ablation and Balloon-atrial-septostomy (CURB) in the Creation of a Stable Inter-atrial Communication:a Preliminary Study in Patients With Pulmonary Arterial Hypertension
Brief Title: Combined Use of Radiofrequency-ablation and Balloon-septostomy in the Creation of a Stable Inter-atrial Communication
Acronym: CURB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-GZ15
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; balloon atrial septostomy; radiofrequency catheter ablation; spontaneous closure
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): Only graded balloon atrial septostomy is carried out, and no radiofrequency catheter ablation is performed.
  Interventions: Other: Balloon atrial septostomy
- single-RFA group (Experimental): After graded balloon atrial septostomy procedure identical to control group, radiofrequency catheter ablation will be performed immediately around the rim of created inter-atrial fenestration.
  Interventions: Other: Radiofrequency catheter ablation; Other: Balloon atrial septostomy
- double-RFA group (Experimental): The first step is radiofrequency catheter ablation on fossae ovalis; and then the other two steps are identical to the single-RFA group (graded balloon atrial septostomy and radiofrequency catheter ablation around the rim of fenestration).
  Interventions: Other: Radiofrequency catheter ablation; Other: Balloon atrial septostomy

INTERVENTIONS:
Other: Radiofrequency catheter ablation — (1) In control group: only graded balloon atrial septostomy will be carried out and there is no radiofrequency catheter ablation. (2) In single-RFA group: after graded balloon atrial septostomy identical to control group, radiofrequency catheter ablation will be performed immediately around the rim of created inter-atrial fenestration. (3) In double-RFA group: the first step is radiofrequency catheter ablation on fossae ovalis; and then the other two steps are identical to the single-RFA group (BAS and RFA around the rim of fenestration).
  Arms: double-RFA group; single-RFA group
Other: Balloon atrial septostomy — Graded balloon atrial septostomy is performed in all patients.

SUMMARY:
Though graded balloon-atrial-septostomy (BAS) has been accepted as an effective palliative therapy for severe pulmonary arterial hypertension, spontaneous closure of septostomy is not uncommon. Radiofrequency-catheter-ablation (RFA), which has the potential to cause irreversible damage around the rim of created inter-atrial communication, might contribute to prevent the spontaneous closure. In patients with severe pulmonary arterial hypertension, the combined use of RFA and BAS (CURB) is investigated to create a stable inter-atrial communication.

DETAILED DESCRIPTION:
Balloon atrial septostomy (BAS) is an important palliative therapy in patients with refractory pulmonary arterial hypertension. However, the incidence of spontaneous closure is higher, which limits the clinical utilization of this procedure. Radiofrequency catheter ablation (RFA) has the potential to cause irreversible damage around the rim of fenestration created with BAS, which might prevent the re-adhesion of the septal remnants. In addition, RFA on fossae ovalis might reduce the elastic recoil of local tissue and contribute to create larger inter-atrial fenestration with same BAS procedure. In this study, the patients between 18 and 60 years of age who have severe pulmonary arterial hypertension associated with right heart failure refractory to medical therapy or severe syncopal symptoms may be eligible for this study (idiopathic severe pulmonary arterial hypertension or severe pulmonary arterial hypertension associated with repaired congenital heart disease). These patients will be randomized 1:1:1 to control group, single-RFA group and double-RFA group:

1. In control group: only BAS is carried out.
2. In single-RFA group: after BAS procedure identical to control group, RFA is performed immediately around the rim of created inter-atrial fenestration.
3. In double-RFA group: the first step is RFA on fossae ovalis; and then the other two steps are identical to the single-RFA group (BAS and RFA around the rim of fenestration).

The immediate size of created fenestration will be determined with intra-cardiac echocardiography, and the patency and size of fenestration will be followed up for 12 months. During the period of follow up, the other evaluations will include the exercise tolerance, cardiac index, systemic arterial oxygen saturation and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic severe pulmonary arterial hypertension;
2. Severe pulmonary arterial hypertension associated with repaired congenital heart disease;
3. World Health Organization functional class III or IV with right heart failure refractory to medical therapy;
4. Severe syncopal symptoms;

Exclusion Criteria:

1. Mean right atrial pressure >20 mm Hg;
2. Room-air resting arterial oxygen saturation <85%;
3. Left ventricular end diastolic pressure (LVEDP) >18mm Hg;
4. Pulmonary vascular resistance >55 wood units/m2.
5. Severe right ventricular failure on cardio-respiratory support
6. The predicted one-year survival <40%;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The size change of the fenestration created with atrial septostomy | 12 months
  The changes of the fenestration-size will be followed up in three different groups

SECONDARY OUTCOMES:
The exercise tolerance | 12 months
  6-min walk test
The systemic arterial oxygen saturation | 12 months
  The change of systemic arterial oxygen saturation after atrial septostomy
World Health Organization functional class | 12 months
  World Health Organization functional class before and after atrial septostomy

CONTACTS AND LOCATIONS:
Overall Officials: Chaowu Yan, PhD and MD, Principal Investigator — National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences,Fuwai Hospital
Locations (1):
- National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences,Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yan C, Wan L, Li H, Wang C, Guo T, Niu H, Li S, Yundan P, Wang L, Fang W. First in-human modified atrial septostomy combining radiofrequency ablation and balloon dilation. Heart. 2022 Oct 13;108(21):1690-1698. doi: 10.1136/heartjnl-2022-321212. PMID 35676068
- [Result] Yan C. Is combined use of radiofrequency ablation and balloon dilation the future of interatrial communications? Expert Rev Cardiovasc Ther. 2022 Nov;20(11):895-903. doi: 10.1080/14779072.2022.2144233. Epub 2022 Nov 10. PMID 36329641